CLINICAL TRIAL: NCT01501227
Title: Comparison of the Incidence of Ventilator Associated Pneumonia in Patients Intubated With the Taper Guard Endotracheal Tube Versus a Normal Endotracheal Tube
Brief Title: Ventilator Associated Pneumonia in Taper Guard Versus Normal Tube in ICU Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Chan Yoo Kuen, Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 859.8
Record Dates: First submitted 2011-12-12; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Ventilator Associated Pneumonia
Keywords: ventilator associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taper Guard Endotracheal Tube (Active Comparator): Patients in the test group will be intubated with the Taper Guard Endotracheal Tube. The incidence of VAP, the length of ventilation, the length of intensive care stay, the length of hospital stay and the mortality rate will be monitored.
  Interventions: Device: Taper Guard Endotracheal Tube
- conventional endotracheal tube (Sham Comparator): Patients in the placebo comparator group will be intubated with the conventional Endotracheal Tube. The incidence of VAP, the length of ventilation, the length of intensive care stay, the length of hospital stay and the mortality rate will be monitored.
  Interventions: Other: Conventional endotracheal tube

INTERVENTIONS:
Device: Taper Guard Endotracheal Tube — comparison of two different endotracheal tubes
  Other Names: Taperguard Evac
  Arms: Taper Guard Endotracheal Tube
Other: Conventional endotracheal tube — Sham Comparator
  Arms: conventional endotracheal tube

SUMMARY:
Ventilator associated pneumonia ( VAP) adds burden to the care of the intensive care patients as they may cause the death of the patient or prolong the intensive care stay or complicate the illness in other ways. The risk of infection is dependent on the interplay between bacteria load into the lungs and the immune status. There has been a lot of focus on bacteria load reduction and this includes the use of subglottic suctioning in an attempt to reduce the amount of bacteria that may move into the lungs. The Hi Lo tubes which were designed to allow subglottic suctioning was significantly effective in reducing the incidence of ventilator associated pneumonia compared to normal tubes. A new generation of endotracheal tubes that not only incorporate subglottic suctioning but provide a more snug fit into the tracheal by a new tapering design may be even more useful to provide the solution for bacterial load reduction. Conventional tubes which may furrow on themselves to allow the creation of microchannels may aid microaspiration. The taper guard which has facilities for subglottic suctioning as well as the strategy to reduce furrowing to the minimum may be the answer to the problem of ventilator associated pneumonia. This study is to determine the extent of protection this tube has against ventilator associated pneumonia compared with conventional endotracheal tubes

DETAILED DESCRIPTION:
Methodology This will be a prospective randomized trial with 2 treatment groups with 100 patients in each arm. The control group ( Group C) will be intubated with our conventional endotracheal tubes and the test group ( Group T) will be intubated with the special Taper guard tubes with subglottic suctioning and snug fit facilities.

All adult patients ( > 18 years of age) admitted into the Intensive Care Unit who are likely to receive more than 72 hours of ventilation will be admitted into the trial. The trial has been cleared by the Hospital Ethics and informed consent will be obtained from the patient's next of kin.

All patients will have their demographic data collected, the primary reason for ICU admission, the APACHE 2 scores, presence of infection at admission, antibiotic use and whether they have risk factors for VAP ( previous surgery, trauma, antibiotics usage, reflux disease and use of stress ulcer prophylaxis, decreased immune status ) The following guidelines modified from the American Thoracic Society 2005 will be used as the basis for diagnosing Ventilator Associated Pneumonia.

Guideline for Diagnosis of Ventilator Associated Pneumonia (VAP)2

1. Patient ventilated for more than 48 hours.
2. Suspicion of ventilation associated pneumonia
3. Presence of a new or progressive infiltrate on chest radiograph.
4. At least 2 of the following:

   1. Fever, defined as an oral temperature greater than 38 degree C, a tympanic temperature greater than 38.5 degree C or a rectal /core temperature greater than 39 degree C OR hypothermia, defined as a rectal/core body temperature of less than 35 degree C.
   2. Elevated total peripheral WBC count (greater than 12000/mm3) or greater than 15% bands regardless of total peripheral WBC count; or leucopenia with total peripheral WBC less than 4500/mm3 (caused by the infection)
   3. New onset of purulent sputum production or other respiratory secretions (e.g. tracheal secretions), or a change in the character of sputum or tracheal secretions
   4. Worsening hypoxaemia with reduction in PaO2/ FiO2 greater or equal to 15%

In addition all patients will have aspirants from the oral cavity (control group) or subglottic region (group T) and the lungs ( both group C and group T) sent on alternate days for bacterial culture. All tubes will be inflated to a sealing pressure of no leak or up to 20-25 cm H2O whichever is the lower.

The sample size has been estimated based on the incidence of ventilation-associated pneumonia (VAP) which is the primary outcome measure from other studies1,2. Based on a VAP incidence of 20% and 6% in each group, 1:1 ratio, 80% power and significance value of 0.05, the number required in each group will be 89. Adding 10% for loss to follow-up, the number needed in each group will be 100 giving a total of 200 The assignment of each patient to the study will be randomized according to computer generated random numbers by the statistician who will not be a party in the ongoing clinical part of the research. In addition she will provide the allocation sequencing via an opaque envelope when a suitable patient has been identified for the assignment of the patient to the 2 groups when informed consent has been obtained. The person who intubates the patient with the endotracheal tube will use the tube that has been allocated according to the written instruction inside the now opened opaque envelope.

Patient and the clinical researchers managing the patient cannot be blinded as there are obvious differences between the 2 types of endotracheal tubes. However the assessor that will determine the presence or absence of the soft signs of ventilator associated pneumonia will be blinded to the type of tubes used. The Radiologist who reads the Chest Xrays will not be privy to the type of tubes used and the Microbiologist determining the significance of the bacteria identified in the oral/subglottic secretions and the tracheal secretions will not be aware of the endotracheal tubes used.

The main outcome measure will be the incidence of ventilator associated pneumonia on each day the patient is ventilated. The secondary outcomes will be the length of ventilation, the duration of intensive care stay, the duration of hospital stay (pre-intensive care, post-intensive care) and the incidence of mortality of the 2 groups.

Statistics Categorical variables will be analysed using Chi square test while continuous variables will be analysed using ANOVA. Intention to treat analysis will be used. Analysis will be carried out using the SPSS version 15.0 software. All statistical tests will be carried out using a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients above 18 years old admitted into the Intensive Care unit and who is to be intubated and likely to receive more than 72 hours of ventilation would be admitted into the trial

Exclusion Criteria:

* presence of cavitary lung disease based on chest x-ray findings,
* primary lung cancer or another metastatic malignancy to the lungs, or known or suspected viral or fungal etiology,
* pneumocystis carinii pneumonia,
* legionella OR Mycoplasma pneumonia or active tuberculosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
incidence of ventilator associated pneumonia(VAP) | 72 hours after ventilation initiated to onset of pneumonia
  the incidence of VAP in patients intubated with the Taper guard tube is compared with the incidence of VAP in patients intubated with the ordinary tube. The criteria for diagnosing VAP is from the American Thoracic Society 2005 guidelines for VAP diagnosis. The assessor for VAP diagnosis is blinded

SECONDARY OUTCOMES:
Number of days on the ventilator by the time patient is discharged from ICU or hospital or at time of death | participants will be followed for the duration of ventilation, an expected average of 2 weeks
  The number of days patient is on the ventilator will be monitored between the 2 groups
The total number of days spent in the intensive care unit by the time of discharge from hospital or death | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  The length of stay in the intensive care unit will be monitored between the 2 groups
The number of days spent in the hospital by the time of discharge or death | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  The length of stay in the hospital will be monitored for the 2 groups
number of deaths in each arm | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  the rate of mortality between the 2 groups will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Kuen Chan, FFARCSI, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, University of Malaya; Vineya Rai, MAnesth; EDIC, Study Director — Department of Anesthesiology, Faculty of Medicine, University of Malaya; Mohd Shahnaz Hassan, MBBS;MAnesth, Study Director — Department of Anesthesiology, Faculty of Medicine, University of Malaya; Suresh Venogobal, MBBS; FANZCA, Study Director — Department of Anesthesiology, Faculty of Medicine, University of Malaya; Kang-Kwong Wong, MBBS;MAnesth, Study Director — Department of Anesthesiology, Faculty of Medicine, University of Malaya; Mohd Yasim Yusof, MBBS;MSc Microbiology, Study Director — Department of Microbiology, Faculty of Medicine, University of Malaya; Foong-Ming Moy, BSc, MSc, MMedSc PH, PhD, Study Director — Julius Centre University of Malaya, Department of Social & Preventive Medicine, Faculty of Medicine, University of Malaya.; Nur Adura Yaakup, MBBS, MRad, Study Director — Department of Biomedical Imaging, Faculty of Medicine, University of Malaya
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Result] Bo H, He L, Qu J. [Influence of the subglottic secretion drainage on the morbidity of ventilator associated pneumonia in mechanically ventilated patients]. Zhonghua Jie He He Hu Xi Za Zhi. 2000 Aug;23(8):472-4. Chinese. PMID 11778260
- [Result] Smulders K, van der Hoeven H, Weers-Pothoff I, Vandenbroucke-Grauls C. A randomized clinical trial of intermittent subglottic secretion drainage in patients receiving mechanical ventilation. Chest. 2002 Mar;121(3):858-62. doi: 10.1378/chest.121.3.858. PMID 11888973
- [Result] Lorente L, Lecuona M, Jimenez A, Mora ML, Sierra A. Influence of an endotracheal tube with polyurethane cuff and subglottic secretion drainage on pneumonia. Am J Respir Crit Care Med. 2007 Dec 1;176(11):1079-83. doi: 10.1164/rccm.200705-761OC. Epub 2007 Sep 13. PMID 17872488
- [Result] Muscedere J, Rewa O, McKechnie K, Jiang X, Laporta D, Heyland DK. Subglottic secretion drainage for the prevention of ventilator-associated pneumonia: a systematic review and meta-analysis. Crit Care Med. 2011 Aug;39(8):1985-91. doi: 10.1097/CCM.0b013e318218a4d9. PMID 21478738